CLINICAL TRIAL: NCT00919698
Title: An Assessment of Delirium in Mechanically Ventilated Patients Undergoing Daily Awakening From Sedation
Brief Title: Delirium in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16938B
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Delirium
Keywords: Hypnotics and Sedatives; Respiration, Artificial; Ventilators, Mechanical; Critical care; Intensive care
MeSH Terms: conditions — Delirium; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sedated mechanically ventilated patients

SUMMARY:
The overall purpose of this trial is to assess the relationship between a daily awakening from sedation and the prevalence of delirium, and in doing so better characterize delirium in the ICU.

DETAILED DESCRIPTION:
This is a single center, observational, cross-over design study assessing the impact of daily awakening from sedation on delirium in the ICU. Enrolled patients will receive a daily baseline delirium assessment using the CAM-ICU tool before the awakening from sedation and an assessment during the awakening from sedation. Each patient will thus serve as their own controls for these interventions.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* intubated and mechanically ventilated
* receiving sedative and/or analgesic medication
* candidate for daily awakening from sedative and/or analgesic medication

Exclusion Criteria:

* primary neurologic disease (stroke, seizure, elevated ICP)
* post cardiac arrest
* do not speak English (assessment only English language validated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (> 18 years old) admitted to the intensive care unit who require mechanical ventilation through an endotracheal tube with infusion of sedative or analgesic medication.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Delirium | Daily

SECONDARY OUTCOMES:
ICU admitting diagnosis | At enrollment
Medications | Daily
Ventilator free days (or first 28) | At 28 days post-intubation
ICU complications | Daily
Days to discharge | At discharge
Survival | At discharge

OTHER OUTCOMES:
survival | 1 year
institution free days | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel SB, Poston JT, Pohlman A, Hall JB, Kress JP. Rapidly reversible, sedation-related delirium versus persistent delirium in the intensive care unit. Am J Respir Crit Care Med. 2014 Mar 15;189(6):658-65. doi: 10.1164/rccm.201310-1815OC. PMID 24423152